CLINICAL TRIAL: NCT03220100
Title: Pilot Study of Stepped Palliative Care in Patients With Advanced Lung Cancer DF/HCC SOCIAL-BEHAVIORAL RESERACH PROTOCOL
Brief Title: Study of Stepped Palliative Care in Patients With Advanced Lung Cancer DF/HCC SOCIAL-BEHAVIORAL RESERACH PROTOCOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Received funding for larger randomized study so terminated pilot study
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jennifer Temel, MD, Director Cancer Outcomes Research, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-284
Record Dates: First submitted 2017-07-10; First posted 2017-07-18 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stepped Palliative Care (Experimental): All participants will receive palliative care Participants will complete the Functional Assessment of Cancer Therapy-Lung (FACT-L) every six weeks FACT-L scores will be used to determine which patients need to step up to every 6 week palliative care visits Patients on step 1 of the intervention will have a palliative care visit every 9 weeks Patients on step 2 of the intervention will have a palliative care visit every 6 weeks
  Interventions: Other: Stepped Palliative Care

INTERVENTIONS:
Other: Stepped Palliative Care — Palliative care clinicians will develop a therapeutic relationship with participants and address their symptoms, coping, prognostic awareness and illness understanding, treatment decision-making, and end of life care needs and preferences.

SUMMARY:
This research study is evaluating a new way to provide palliative care to patients who have recently been diagnosed with lung cancer. . Palliative care is a medical specialty focused on lessening (or "palliating") patients' symptoms and helping patients and their families cope with a serious illness.

DETAILED DESCRIPTION:
Patients with serious cancers, like advanced lung cancer, often experience physical symptoms, such as pain or shortness of breath. Both patients and their families often feel worried and/or sad about this diagnosis. Research has shown that early involvement of a team of clinicians that specialize in lessening (or palliating) many of these distressing physical and emotional symptoms, and in helping patients and their families' cope with serious illnesses, improves patients' quality of life and mood, and can help their loved ones' feel less depressed or sad. This team is called "palliative care," and consists of physicians and advanced practice nurses who work closely and collaboratively with the oncology team to care for the patient and their loved ones.

While the investigators know having palliative care clinicians care for patients along with their oncology team is helpful for the participant and their loved ones, the investigators do not know the optimal timing of the visits with palliative care.

The purpose of this study is to see if the investigators can closely monitor participants' health condition and quality of life and use these metrics as indications of when the participant should see the palliative care team.

This study will monitor participants' health condition and schedule the participant to see the palliative care team if the participants' cancer grows or after the participant have been admitted to the hospital. The investigators will also monitor participants' quality of life every six weeks and schedule the participant to see the palliative care monthly if the participant quality of life decreases during the study.

This study will also monitor participants' mood, coping, and understanding of the participant illness and prognosis. The investigators will ask the participant to fill out questionnaires asking about these topics every 12 weeks. The participant will be able to complete these questionnaires in clinic, via email, using a mailed paper copy, or over the phone with a member of the research team.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with advanced non-small cell lung cancer, small cell lung cancer, or mesothelioma, being treated with non-curative intent, and informed of advanced disease within the prior eight weeks
* Eastern Cooperative Oncology Group (ECOG) Performance Status from 0 (asymptomatic) to 2 (symptomatic and in bed <50% of the day)
* The ability to read and respond to questions in English or with minimal help from a family member or medical interpreter.
* Primary cancer care at the MGH Cancer Center
* Age > 18 years

Exclusion Criteria:

* They are already receiving PC or hospice services
* They have cognitive or psychiatric conditions as determined by the treating oncologist that prohibits study consent or participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who complete the study protocol | 2 years
  The investigators will determine that the study protocol is feasible if at least 75% of participants on step 2 of the intervention complete at least 70% of the scheduled palliative care visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Temel, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No